CLINICAL TRIAL: NCT00400725
Title: Comparison of the Maintenance Effect of Clobex® Shampoo 0.05% Used Twice Weekly vs. Vehicle on Scalp Psoriasis in Subjects Who Successfully Responded to a 4-week Daily Course of Clobex® Shampoo 0.05%
Brief Title: Maintenance Effect of Clobex Shampoo on Participants With Moderate to Severe Scalp Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RD.03.SPR.29060
Record Dates: First submitted 2006-11-16; First posted 2006-11-17 (Estimated); Results first posted 2023-07-11 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2022-08

CONDITIONS: Scalp Psoriasis
Keywords: maintenance; scalp psoriasis; Galderma
MeSH Terms: interventions — Clobetasol

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Initial Phase:- Clobex® Shampoo (Experimental): In initial open-label phase, participants were applied Clobex® shampoo (Clobetasol Propionate) 0.05 percent (%) weight by weight (W/W) topically to the scalp once daily (twice a week) for 4 weeks (weekly dose was not more than 50 grams [50 Milliliter]).
  Interventions: Drug: Clobex® Shampoo
- Maintenance Phase: Clobex® Shampoo (Experimental): In maintenance double-blind phase, participants presented with a good efficacy (Global severity score [GSS] less than or equal to [<=] 2) in initial phase were randomized to apply Clobetasol Propionate shampoo 0.05 % weight by weight (W/W) twice weekly up to 6 months (wherein weekly dose were not exceeded beyond 50 grams [50 milliliter]). In case of relapse (that is [i.e.], GSS greater than [>] 2) participants were re-entered to 4-week daily treatment with Clobetasol Propionate shampoo 0.05%. After this 4-week period of daily treatment, if GSS <= 2, participants were re-entering the maintenance regimen (twice a week).
  Interventions: Drug: Clobex® Shampoo
- Maintenance Phase: Clobex® Vehicle Shampoo (Placebo Comparator): In maintenance double-blind phase, participants presented with a good efficacy (Global severity score [GSS] <= 2) in initial phase were randomized to apply Clobex® vehicle shampoo twice weekly up to 6 months (wherein weekly dose was not more than 50 grams [50 milliliter]). In case of relapse (i.e., GSS [greater than] > 2) participants were re-entered to 4-week daily treatment with Clobetasol Propionate Shampoo 0.05 % (W/W). After this 4-week period of daily treatment, if GSS <= 2, participants were re-entering the maintenance regimen (twice a week).
  Interventions: Drug: Clobex® Vehicle Shampoo

INTERVENTIONS:
Drug: Clobex® Shampoo — Clobex® Shampoo 0.05 % (W/W) topically to scalp for 4 weeks.
  Other Names: Clobetasol Propionate 0.05% [weight by weight (W/W)]
  Arms: Initial Phase:- Clobex® Shampoo
Drug: Clobex® Vehicle Shampoo — Clobex® Vehicle Shampoo 0.05 % (W/W) topically to scalp up to 6 months.
  Arms: Maintenance Phase: Clobex® Vehicle Shampoo
Drug: Clobex® Shampoo — Clobex® Shampoo 0.05% (W/W) topically to scalp up to 6 months.
  Other Names: Clobetasol Propionate 0.05% (W/W)
  Arms: Maintenance Phase: Clobex® Shampoo

SUMMARY:
The objective of the study was to assess the maintenance effect on scalp psoriasis of Clobex® Shampoo 0.05% when used twice weekly.

DETAILED DESCRIPTION:
Psoriasis was a chronic disease that was affecting skin, the scalp and joints. Scalp psoriasis was very common and was having an important impact on people's life.

Primary objective of scalp psoriasis treatments was to gain initial and rapid control of the disease process with a minimum of side-effects and improve patient quality of life.

Still, one of the unmet needs of scalp psoriasis therapies was the maintenance of a long-term remission. For corticosteroids in particular, one of the drawbacks was the disease recurrences after cessation of the treatment.

Therefore, the establishment of a modified corticosteroid dosing regimen that would allow remission with minimal side-effects was suitable.

The purpose of this study was to assess how long a patient successfully maintained in a good condition after use of Clobex® shampoo only twice a week.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 18 years or older.
* Subjects with moderate to severe scalp psoriasis

Exclusion Criteria:

* Subjects who needed systemic treatment for their body psoriasis
* Subjects with a washout period for topical treatment(s) on the scalp less than:

  * Corticosteroids 2 weeks
  * All other anti-psoriasis medications 2 weeks
* Subjects with a washout period for systemic treatment(s) less than:

  * PUVA therapy 4 weeks
  * Biological therapies 12 weeks
  * Treatments other than biologicals with a possible efficacy on psoriasis 4 weeks
  * Treatment known to worsen psoriasis 2 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2006-09-29 (Actual); Primary Completion 2007-08-20 (Actual); Study Completion 2007-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Poulin, MD, Principal Investigator — Centre de Recherche Dermatologique du Quebec Métropolitain
Locations (1):
- centre de Recherche Dermatologique du Québec, Québec, Canada

REFERENCES:
- See also: Related Info — http://www.clobex.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 12 sites in Canada from 29 September 2006 (first participant first visit) to 20 August 2007 (last participant last visit).
Pre-assignment Details: A total of 288 participants were enrolled in initial phase of the study, of which 225 participants were eligible to enter maintenance phase after completion of initial phase. Out of 225 eligible participants, only 217 participants (as 8 participants withdrew consent) were randomized and received treatment in the maintenance phase either in Clobetasol Propionate Shampoo group or Vehicle group.
Groups:
- Initial Phase:- Clobex® Shampoo: In initial open-label phase, participants were applied Clobetasol Propionate shampoo 0.05 percent (%) weight by weight (W/W) topically to the scalp once daily (twice a week) for 4 weeks (weekly dose was not more than 50 grams [50 Milliliter]).
- Maintenance Phase: Clobex® Shampoo: In maintenance double-blind phase, participants presented with a good efficacy (Global severity score [GSS] less than or equal to [<=] 2) in initial phase were randomized to apply Clobetasol Propionate shampoo 0.05 percent (%) weight by weight (W/W) twice weekly up to 6 months (wherein weekly dose were not exceeded beyond 50 grams [50 milliliter]). In case of relapse (that is [i.e.], GSS greater than [>] 2) participants were re-entered to 4-week daily treatment with Clobetasol Propionate shampoo 0.05%. After this 4-week period of daily treatment, if GSS <= 2, participants were re-entering the maintenance regimen (twice a week).
- Maintenance Phase:Clobex® Vehicle Shampoo: In maintenance double-blind phase, participants presented with a good efficacy (Global severity score [GSS] <= 2) in initial phase were randomized to apply Clobex® vehicle shampoo twice weekly up to 6 months (wherein weekly dose were not exceeded beyond 50 grams [50 milliliter]). In case of relapse (that is [i.e.], GSS [greater than] > 2) participants were re-entered to 4-week daily treatment with Clobetasol Propionate Shampoo 0.05 percent (%) weight by weight (W/W). After this 4-week period of daily treatment, if GSS <= 2, participants were re-entering the maintenance regimen (twice a week).
Period: Initial Phase (up to 4 Weeks)
Arm/Group | Initial Phase:- Clobex® Shampoo | Maintenance Phase: Clobex® Shampoo | Maintenance Phase:Clobex® Vehicle Shampoo
Started | 288 | 0 | 0
Completed | 271 | 0 | 0
Not Completed | 17 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Withdrawal by Subject | 14 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Other | 1 | 0 | 0
Period: Maintenance Phase (up to 6 Months)
Arm/Group | Initial Phase:- Clobex® Shampoo | Maintenance Phase: Clobex® Shampoo | Maintenance Phase:Clobex® Vehicle Shampoo
Started | 0 | 106 (271 participants completed initial phase, of which 217 participants were randomized to the maintenance phase.) | 111 (271 participants completed initial phase, of which 217 participants were randomized to the maintenance phase)
Completed | 0 | 90 | 82
Not Completed | 0 | 16 | 29
Not completed — Lack of Efficacy | 0 | 1 | 0
Not completed — Adverse Event | 0 | 2 | 4
Not completed — Withdrawal by Subject | 0 | 11 | 21
Not completed — Lost to Follow-up | 0 | 1 | 2
Not completed — Other | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Population: ITT Population included the entire population who were enrolled and randomized. (i.e., assigned a kit number). As per planned analysis, baseline data for all participants were collected at initial phase only.
Groups:
- All Participants: In initial open-label phase, participants were applied Clobetasol Propionate shampoo 0.05% topically to the scalp once daily (twice a week) for 4 weeks (wherein weekly dose was not more than 50 grams [50 milliliter]). In maintenance double-blind phase, participants presented with a good efficacy (GSS <= 2) in initial phase were randomized to apply Clobetasol Propionate Shampoo 0.05% (W/W) or Clobex® Vehicle Shampoo twice weekly up to 6 months (wherein weekly dose was not more than 50 grams [50 milliliter]). In case of relapse (i.e., GSS > 2) participants were re-entered to 4-week daily treatment with Clobetasol Propionate Shampoo 0.05%. After this 4-week period of daily treatment, if GSS <= 2, participants were re-entering the maintenance regimen (twice a week).
Arm/Group | All Participants
Number analyzed (Participants) | 288
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.4 (16.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 166
  Male | 122
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasian | 265
  Race: Black | 1
  Race: Asian | 13
  Race: Hispanic | 6
  Race: Other | 3

OUTCOME MEASURES:

1. Primary Outcome: Maintenance Phase: Time to First Relapse
Description: Time to first relapse was defined as the duration between baseline of maintenance phase and the visit where the relapse occurred. The first relapse was defined as the first time during the maintenance phase when participant presented with a GSS >2.
Time Frame: Baseline up to 24 Weeks
Population: ITT Population included the entire population who were enrolled and randomized (i.e., assigned a kit number).
Measure: Mean (Standard Error); unit: days
Groups:
- Maintenance Phase: Clobex® Shampoo: In maintenance double-blind phase, participants presented with a good efficacy (GSS <=2) in initial phase were randomized to apply Clobetasol Propionate shampoo 0.05% (W/W) twice weekly up to 6 months (wherein weekly dose was not more than 50 grams [50 milliliter]). In case of relapse (i.e., GSS > 2) participants were re-entered to 4-week daily treatment with Clobetasol Propionate shampoo 0.05% (W/W). After this 4-week period of daily treatment, if GSS <= 2, participants were re-entering the maintenance regimen (twice a week).
- Maintenance Phase: Clobex® Vehicle Shampoo: In maintenance double-blind phase, participants presented with a good efficacy (GSS <=2) in initial phase were randomized to apply Clobex® vehicle shampoo twice weekly up to 6 months (wherein weekly dose was not more than 50 grams [50 milliliter]). In case of relapse (i.e., GSS > 2) participants were re-entered to 4-week daily treatment with Clobetasol Propionate Shampoo 0.05% (W/W). After this 4-week period of daily treatment, if GSS <= 2, participants were re-entering the maintenance regimen (twice a week).
Arm/Group | Maintenance Phase: Clobex® Shampoo | Maintenance Phase: Clobex® Vehicle Shampoo
Number analyzed (Participants) | 106 | 111
days | 93.5 (6.5) | 56.8 (4.7)

2. Secondary Outcome: Initial Phase: Percentage of Participants With Global Severity Scores
Description: Global severity score was evaluated on a scale of 0-4 and it was categorized as; Clear (score 0); no clinical signs or symptoms detected (hyperpigmentation or residual red coloration might be present), very mild (score 1); only very slight signs or symptoms detected (e.g., very fine scaling or slight erythema), mild (score 2); slight signs or symptoms detected (e.g., mild erythema and scaling, eventually associated to some barely detectable plaque elevation), moderate (score 3); moderate or clearly detectable signs or symptoms (e.g., definite redness with obvious scaling on a plaque that was elevated above skin level), severe (score 4); severe signs or symptoms detected (e.g., intense redness, profuse shedding, definite plaque thickness was most often present) where 0 indicates best and 4 indicates worst. Percentage of participants with GSS was reported. Missing Clobex® shampoo data were imputed using last observation carried forward (LOCF).
Time Frame: Baseline, Weeks 2 and 4 LOCF
Population: ITT Population included the entire population who were enrolled and randomized. (i.e., assigned a kit number).
Measure: Number; unit: percentage of participants
Groups:
- Initial Phase:- Clobex® Shampoo (Clobetasol Propionate 0.05% [W/W]): In initial open-label phase, participants were applied Clobetasol Propionate 0.05% (W/W) shampoo topically to the scalp once daily (twice a week) for 4 weeks (weekly dose was not more than 50 grams [50 Milliliter]).
Arm/Group | Initial Phase:- Clobex® Shampoo (Clobetasol Propionate 0.05% [W/W])
Number analyzed (Participants) | 288
percentage of participants
  Baseline: Score 0 (Clear) | 0
  Baseline: Score 1 (Very mild) | 0
  Baseline: Score 2 (Mild) | 0
  Baseline: Score 3 (Moderate) | 58.3
  Baseline: Score 4 (Severe) | 41.7
  Week 2-LOCF: Score 0 (Clear) | 2.4
  Week 2-LOCF: Score 1 (Very mild) | 10.1
  Week 2-LOCF: Score 2 (Mild) | 35.4
  Week 2-LOCF: Score 3 (Moderate) | 43.1
  Week 2-LOCF: Score 4 (Severe) | 9.0
  Week 4-LOCF: Score 0 (Clear) | 7.6
  Week 4-LOCF: Score 1 (Very mild) | 25.3
  Week 4-LOCF: Score 2 (Mild) | 45.1
  Week 4-LOCF: Score 3 (Moderate) | 18.4
  Week 4-LOCF: Score 4 (Severe) | 3.5

3. Secondary Outcome: Initial Phase: Percentage of Participants With Pruritus Scores
Description: Pruritus (itching sensation) score of were evaluated on a scale from 0 - 3 (0 = None [no itching], 1 = Mild [slight itching], not really bothersome), 2 = Moderate [definite itching that is somewhat bothersome; without loss of sleep], and 3 = severe [intense itching that has caused pronounced discomfort; night rest interrupted and excoriations of the skin from scratching may be present]) , where 0 indicates best and 3 indicates worst. Percentage of participants with pruritus score was reported. Missing Clobex® shampoo data were imputed using last observation carried forward (LOCF).
Time Frame: Baseline, Weeks 2 and 4 LOCF
Population: ITT Population included the entire population who were enrolled and randomized. (i.e., assigned a kit number).
Measure: Number; unit: percentage of participants
Groups:
- Initial Phase:- Clobex® Shampoo: In initial open-label phase, participants were applied Clobetasol Propionate 0.05% (W/W) shampoo topically to the scalp once daily (twice a week) for 4 weeks (weekly dose was not more than 50 grams [50 Milliliter]).
Arm/Group | Initial Phase:- Clobex® Shampoo
Number analyzed (Participants) | 288
percentage of participants
  Baseline: Score 0 (None) | 3.8
  Baseline: Score 1 (Mild) | 20.8
  Baseline: Score 2 (Moderate) | 51.7
  Baseline: Score 3 (Severe) | 23.6
  Week 2- LOCF: Score 0 (None) | 19.8
  Week 2- LOCF: Score 1 (Mild) | 53.5
  Week 2- LOCF: Score 2 (Moderate) | 23.6
  Week 2- LOCF: Score 3 (Severe) | 3.1
  Week 4- LOCF: Score 0 (None) | 35.4
  Week 4- LOCF: Score 1 (Mild) | 47.6
  Week 4- LOCF: Score 2 (Moderate) | 15.6
  Week 4- LOCF: Score 3 (Severe) | 1.4

4. Secondary Outcome: Initial Phase: Percentage of Participants With Individual Category of Scalp Psoriasis Individual Signs (Erythema, Scaling and Plaque Thickening) Scores
Description: Individual sign scores of erythema (abnormal redness of skin), scaling (scales attached to the scalp), plaque thickening (a thickening or elevation of a circumscribed lesion or plaque) were evaluated on a scale of 0-4; 0= none , 1= mild , 2=moderate , 3= severe, 4= very severe, where 0 indicates best and 4 indicates worst. Percentage of participants with individual signs (erythema, scaling, and plaque thickening) scores were reported. Missing Clobex® shampoo data were imputed using last observation carried forward (LOCF).
Time Frame: Baseline, Weeks 2 and 4 LOCF
Population: ITT Population included the entire population who were enrolled and randomized. (i.e., assigned a kit number).
Measure: Number; unit: percentage of participants
Arm/Group | Initial Phase:- Clobex® Shampoo
Number analyzed (Participants) | 288
percentage of participants
  Erythema at Baseline: Score 0 (None) | 0
  Erythema at Baseline: Score 1 (Mild) | 1.7
  Erythema at Baseline: Score 2 (Moderate) | 47.2
  Erythema at Baseline: Score 3 (Severe) | 45.5
  Erythema at Baseline: Score 4 (Very Severe) | 5.6
  Erythema at Week 2 - LOCF: Score 0 (None) | 2.4
  Erythema at Week 2 - LOCF: Score 1 (Mild) | 39.6
  Erythema at Week 2 - LOCF : 2: Moderate | 44.1
  Erythema at Week 2 - LOCF: Score 3 (Severe) | 13.2
  Erythema at Week 2 - LOCF: Score 4 (Very Severe) | 0.4
  Erythema at Week 4 - LOCF: Score 0 (None) | 12.2
  Erythema at Week 4 - LOCF: Score 1 (Mild) | 51.4
  Erythema at Week 4 - LOCF: Score 2 (Moderate) | 30.9
  Erythema at Week 4 - LOCF: Score 3 (Severe) | 4.9
  Erythema at Week 4 - LOCF: Score 4 (Very Severe) | 0.7
  Scaling at Baseline: Score 0 (None) | 0
  Scaling at Baseline: Score 1 (Mild) | 0.7
  Scaling at Baseline: Score 2 (Moderate) | 42.0
  Scaling at Baseline: Score 3 (Severe) | 49.7
  Scaling at Baseline: Score 4: (Very Severe) | 7.6
  Scaling at Week 2-LOCF: Score 0 (None) | 5.9
  Scaling at Week 2-LOCF: Score 1 (Mild) | 35.1
  Scaling at Week 2-LOCF: Score 2 (Moderate) | 45.5
  Scaling at Week 2-LOCF: Score 3 (Severe) | 10.8
  Scaling at Week 2-LOCF: Score 4 (Very Severe) | 2.8
  Scaling at Week 4-LOCF: Score 0 (None) | 14.2
  Scaling at Week 4-LOCF: Score 1 (Mild) | 50.7
  Scaling at Week 4-LOCF: Score 2 (Moderate) | 30.6
  Scaling at Week 4-LOCF: Score 3 (Severe) | 3.5
  Scaling at Week 4-LOCF: Score 4 (Very Severe) | 1.0
  Plaque Thickening at Baseline: Score 0 (None) | 0.7
  Plaque Thickening at Baseline: score 1 (Mild) | 4.9
  Plaque Thickening at Baseline: Score 2 (Moderate) | 54.2
  Plaque Thickening at Baseline: Score 3 (Severe) | 36.5
  Plaque Thickening at Baseline: Score 4 (Very Severe) | 3.8
  Plaque Thickening at Week 2-LOCF: Score 0 (None) | 10.8
  Plaque Thickening at Week 2-LOCF: Score 1 (Mild) | 37.5
  Plaque Thickening at Week 2-LOCF: Score 2 (Moderate) | 43.4
  Plaque Thickening at Week 2-LOCF: Score 3 (Severe) | 6.9
  Plaque Thickening at Week 2- LOCF: Score 4 (Very Severe) | 1.4
  Plaque Thickening at Week 4- LOCF: Score 0 (None) | 23.6
  Plaque Thickening at Week 4- LOCF: Score 1 (Mild) | 49.3
  Plaque Thickening at Week 4-LOCF: Score 2 (Moderate) | 23.3
  Plaque Thickening at Week 4- LOCF: Score 3 (Severe) | 2.8
  Plaque Thickening at Week 4- LOCF: Score 4 (Very Severe) | 1.0

5. Secondary Outcome: Maintenance Phase: Percentage of Participants Who Had First Relapse
Description: The first relapse was defined as the first time during the maintenance phase when participant presented with a GSS >2. Relapse was categorized into relapse or no relapse. Percentage of participants with relapse were reported.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: ITT worstcase population signifies participants who prematurely discontinued before the time of first relapse were considered as relapse at following visit. Here, "number analyzed" refer to participants evaluable for this outcome at given timepoints.
Measure: Number; unit: percentage of participants
Groups:
- Maintenance Phase: Clobex® Shampoo: In maintenance double-blind phase, participants presented with a good efficacy (GSS <= 2) in initial phase (i.e., last initial phase visit [maintenance baseline]) were randomized to apply Clobetasol Propionate shampoo 0.05% (W/W) twice weekly up to 6 months (wherein weekly dose was not more than 50 grams [50 milliliter]). In case of relapse [i.e., GSS > 2] participants were re-entered to 4-week daily treatment with Clobetasol Propionate shampoo 0.05% (W/W). After this 4-week period of daily treatment, if GSS <= 2, participants were re-entering the maintenance regimen (twice a week).
- Maintenance Phase: Clobex® Vehicle Shampoo: In maintenance double-blind phase, participants presented with a good efficacy (GSS ≤ 2) in initial phase were randomized to apply Clobex® vehicle shampoo twice weekly up to 6 months (wherein weekly dose was not more than 50 grams [50 milliliter]). In case of relapse (i.e., GSS > 2) participants were re-entered to 4-week daily treatment with Clobetasol Propionate shampoo 0.05% (W/W). After this 4-week period of daily treatment, if GSS <= 2, participants were re-entering the maintenance regimen (twice a week).
Arm/Group | Maintenance Phase: Clobex® Shampoo | Maintenance Phase: Clobex® Vehicle Shampoo
Number analyzed (Participants) | 106 | 111
percentage of participants
  Maintenance Baseline : Relapse | 0 | 0
  Week 4 : Relapse: number analyzed (Participants) | 105 | 110
  Week 4 : Relapse | 41 | 64.5
  Week 8 : Relapse | 52.8 | 76.6
  Week 12 : Relapse: number analyzed (Participants) | 106 | 110
  Week 12 : Relapse | 55.7 | 84.5
  Week 16 : Relapse: number analyzed (Participants) | 105 | 111
  Week 16 : Relapse | 62.9 | 89.2
  Week 20 : Relapse: number analyzed (Participants) | 105 | 111
  Week 20 : Relapse | 66.7 | 90.1
  Week 24 : Relapse | 68.9 | 91.9

6. Secondary Outcome: Maintenance Phase: Percentage of Participants With Scalp Psoriasis Pruritus Score at First Time of Relapse
Description: Pruritus (itching sensation) score of were evaluated on a scale from 0 - 3 (0 = None [no itching], 1 = Mild [slight itching, not really bothersome], 2 = Moderate [definite itching that is somewhat bothersome; without loss of sleep], and 3 = severe [intense itching that has caused pronounced discomfort; night rest interrupted and excoriations of the skin from scratching may be present]) , where 0 indicates best and 3 indicates worst. Percentage of participants with scalp psoriasis pruritus score at first relapse was reported.
Time Frame: Baseline up to Week 24
Population: ITT worstcase population signifies participants who prematurely discontinued before the time of first relapse were considered as relapse at following visit. Overall number of participants analyzed refer to the participants evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Groups:
- Maintenance Phase: Clobex® Shampoo: In maintenance double-blind phase, participants presented with a good efficacy (GSS <= 2) in initial phase were randomized to apply Clobetasol Propionate shampoo 0.05% (W/W) twice weekly up to 6 months (wherein weekly dose was not more than 50 grams [50 milliliter]). In case of relapse [i.e., GSS > 2] participants were re-entered to 4-week daily treatment with Clobetasol Propionate shampoo 0.05% (W/W). After this 4-week period of daily treatment, if GSS <= 2, participants were re-entering the maintenance regimen (twice a week).
Arm/Group | Maintenance Phase: Clobex® Shampoo | Maintenance Phase: Clobex® Vehicle Shampoo
Number analyzed (Participants) | 68 | 97
percentage of participants
  0: None | 13.2 | 7.2
  1: Mild | 29.4 | 26.8
  2: Moderate | 51.5 | 52.6
  3: Severe | 5.9 | 13.4

7. Secondary Outcome: Maintenance Phase: Percentage of Participants With Individual Category of Scalp Psoriasis Individual Signs (Erythema, Scaling and Plaque Thickening) Scores at First Time of Relapse
Description: The first relapse was defined as the first time during the maintenance phase when participant presented with a GSS >2. Individual sign scores of erythema were evaluated on a scale of 0-4 (0= none, 1= mild, 2=moderate, 3= severe, 4= very severe), where 0 indicates best and 4 indicates worst. Percentage of participants with individual signs (erythema, scaling and plaque thickening) scores were reported. There were no participants in scaling category with 0 score.
Time Frame: Baseline up to Week 24
Population: ITT Population included the entire population who were enrolled and randomized (i.e., assigned a kit number). Here, overall number of participants analyzed refer to the participants evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Maintenance Phase: Clobex® Shampoo | Maintenance Phase: Clobex® Vehicle Shampoo
Number analyzed (Participants) | 68 | 97
percentage of participants
  Erythema: Score 0 (None) | 1.5 | 0
  Erythema: Score 1 (Mild) | 13.2 | 13.4
  Erythema: Score 2 (Moderate) | 57.4 | 54.6
  Erythema: Score 3 (Severe) | 25.0 | 30.9
  Erythema: Score 4 (Very Severe) | 2.9 | 1
  Scaling: Score 1 (Mild) | 4.4 | 4.1
  Scaling: Score 2 (Moderate) | 57.4 | 64.9
  Scaling: Score 3 (Severe) | 35.3 | 29.9
  Scaling: Score 4 (Very Severe) | 2.9 | 1.0
  Plaque Thickening: Score 0 (None) | 1.5 | 2.1
  Plaque Thickening: Score 1 (Mild) | 17.6 | 14.4
  Plaque Thickening: Score 2 (Moderate) | 64.7 | 67.0
  Plaque Thickening : Score 3 (Severe) | 16.2 | 14.4
  Plaque Thickening: Score 4 (Very Severe) | 0 | 2.1

8. Secondary Outcome: Maintenance Phase: Percentage of Participants With Number of Relapses Experienced
Description: Number of relapses of participants were categorized as 0; zero relapse, 1; one relapse, 2; two relapse, 3; three relapse, 4; two consecutive relapses.
  Percentage of participants with total number of relapses experienced during maintenance period was reported.
Time Frame: Baseline up to Week 28
Population: ITT worstcase population signifies participants who prematurely discontinued before the time of first relapse were considered as relapse at following visit.
Measure: Number; unit: percentage of participants
Groups:
- Clobex® Shampoo: In maintenance double-blind phase, participants presented with a good efficacy (GSS <= 2) in initial phase were randomized to apply Clobetasol Propionate shampoo 0.05% (W/W) twice weekly up to 6 months (wherein weekly dose was not more than 50 grams [50 milliliter]). In case of relapse [i.e., GSS > 2] participants were re-entered to 4-week daily treatment with Clobetasol Propionate shampoo 0.05% (W/W). After this 4-week period of daily treatment, if GSS <= 2, participants were re-entering the maintenance regimen (twice a week).
- Clobex® Vehicle Shampoo: In maintenance double-blind phase, participants presented with a good efficacy (GSS ≤ 2) in initial phase were randomized to apply Clobex® vehicle shampoo twice weekly up to 6 months (wherein weekly dose was not more than 50 grams [50 milliliter]). In case of relapse (i.e., GSS > 2) participants were re-entered to 4-week daily treatment with Clobetasol Propionate shampoo 0.05% (W/W). After this 4-week period of daily treatment, if GSS <= 2, participants were re-entering the maintenance regimen (twice a week).
Arm/Group | Clobex® Shampoo | Clobex® Vehicle Shampoo
Number analyzed (Participants) | 106 | 111
percentage of participants
  0: Zero Relapse | 31.1 | 8.1
  1: One Relapse | 26.4 | 22.5
  2: Two Relapse | 9.4 | 25.2
  3: Three Relapse | 7.5 | 18.0
  4: Two Consecutive Relapses | 25.5 | 26.1

ADVERSE EVENTS:
Time Frame: From baseline up to Week 28
Description: Analysis was performed on safety population that included in the study. Safety population was defined as intent-to-treat population (entire population enrolled and randomized i.e., assigned a kit number), after exclusion of participants who never applied treatment with certainty based on monitoring report.
Arm/Group | Initial Phase:- Clobex® Shampoo | Maintenance Phase: Clobex® Shampoo | Maintenance Phase: Clobex® Vehicle Shampoo
All-Cause Mortality (participants affected / at risk) | 1/288 | 0/106 | 0/111
Serious Adverse Events (participants affected / at risk) | 3/288 | 2/106 | 5/111
Other Adverse Events (participants affected / at risk) | 39/288 | 44/106 | 45/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Initial Phase:- Clobex® Shampoo (N=288) | Maintenance Phase: Clobex® Shampoo (N=106) | Maintenance Phase: Clobex® Vehicle Shampoo (N=111)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Aortic aneurysm rupture (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Renal cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Abdominal Hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Initial Phase:- Clobex® Shampoo (N=288) | Maintenance Phase: Clobex® Shampoo (N=106) | Maintenance Phase: Clobex® Vehicle Shampoo (N=111)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 2 (2) | 2 (2) | 6 (6)
Gastroesophageal reflux Disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Colitis Ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (5)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Inguinal Hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Influenza Like Illness (General disorders) | 1 (1) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1)
Odema Peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis Viral (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 1 (1) | 5 (5)
Lice Infestation (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nesopharyngitis (Infections and infestations) | 12 (12) | 10 (12) | 10 (11)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0) | 1 (2)
Upper Respiratory Tract Infection (Infections and infestations) | 3 (3) | 4 (4) | 4 (4)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Chronic Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Otitis Externa (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Otitis Media (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Streptococcal Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Vaginal Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tendon Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Back Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Foot Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Foreign Body in eye (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Muscle Strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Post-traumatic Pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram Abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood Cortisol Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Psoriatic Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (3)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hair Colour Changes (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Skin Burning Sensation (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1) | 1 (1)
Skin Discomfort (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Folliculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Hypotrichosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Tinea Versicolour (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dermal Cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Cardiac Flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Angina Pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Urinary Incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Hysterectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Dental Prosthesis Placement (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal Dryness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 4 (5)
Transient Ischemic Attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other